CLINICAL TRIAL: NCT01545843
Title: Repeated Partial Sleep Deprivation to Augment SSRI Response in Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, J. Todd Arnedt, Assistant Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH077690 (NIH)
Record Dates: First submitted 2012-01-12; First posted 2012-03-07 (Estimated); Results first posted 2015-01-30 (Estimated); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Depression
Keywords: depression; sleep; treatment
MeSH Terms: conditions — Depression | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- No sleep deprivation (Active Comparator): Sleep scheduling plus fluoxetine. 8 hours time in bed for two weeks plus fluoxetine for 8 weeks
  Interventions: Behavioral: Sleep scheduling; Drug: Fluoxetine
- Late bedtime sleep deprivation (Experimental): Sleep scheduling plus fluoxetine. 6 hours time in bed for two weeks plus fluoxetine for 8 weeks. Bedtime delayed by 2 hours.
  Interventions: Behavioral: Sleep scheduling; Drug: Fluoxetine
- Early risetime sleep deprivation (Experimental): Sleep scheduling plus fluoxetine. 6 hours time in bed for two weeks plus fluoxetine for 8 weeks. Risetime advanced by 2 hours.
  Interventions: Behavioral: Sleep scheduling; Drug: Fluoxetine

INTERVENTIONS:
Behavioral: Sleep scheduling — 8 hours vs. 6 hours time in bed for two weeks, with either 2 hour advance of risetime, or 2 hour delay of bedtime
Drug: Fluoxetine — 20-40 mg fluoxetine daily for 8 weeks
  Other Names: Prozac

SUMMARY:
The purpose of the study is to determine whether changing sleep patterns improves response to an antidepressant medication.

DETAILED DESCRIPTION:
Depression is common and associated with social and economic costs. Although antidepressant medications are an effective treatment for depression, it can take as long as 6-8 weeks before symptoms improve, and 20-35% of individuals who use antidepressants still experience depression symptoms.

New treatments that accelerate response to antidepressants are important to reduce the burden of depression. The objectives of the proposed study are (1) to evaluate the effects of partial sleep deprivation compared to no sleep deprivation for improving response to 8 weeks of fluoxetine 20-40 mg treatment and (2) to examine the underlying sleep mechanisms of treatment response.

Participants who are eligible for the study will be randomly assigned to one of three sleep schedules for a 2-week period while taking fluoxetine: no sleep deprivation (8 hours time in bed), late bedtime (6 hours time in bed, with 2 hour bedtime delay) or early risetime (6 hours time in bed, with 2 hour advancement of rise time). Participants will spend a total of 7 nights in our sleep laboratory and will be followed on fluoxetine for an 8-week period.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years old
* Current major depressive episode
* Habitual TIB of 7 to < 10 hours
* No antidepressant medications for ≥ 2 weeks (4 weeks for MAOIs or longer acting antidepressants)
* Score of at least 18 on the Hamilton Rating Scale of Depression

Exclusion Criteria:

* Alcohol or substance abuse/dependence in past 6 months
* Current posttraumatic stress disorder or bulimia nervosa (past 6 months)
* Lifetime history of bipolar I or II disorder, schizophrenia/other psychotic disorder, and anorexia nervosa
* Trials of fluoxetine in the past 6 months
* Medical disorders or pain syndromes that may affect sleep or are associated with significant depression (e.g. thyroid or Cushing's disease); history of head trauma with loss of consciousness of > 5 minutes; history of seizures
* Sleep disorders other than insomnia, such as sleep apnea and periodic limb movement disorder
* Current use of prescription, over-the-counter, or naturopathic remedies for sleep (e.g., barbiturates, benzodiazepine agonists, nonbenzodiazepine hypnotics, analgesics) or depression (e.g., Sam-E, St. John's Wort)
* Currently working evening or midnight shift (subjects who have recently traveled across multiple time zones will be included at the discretion of the PI).
* Currently at risk for drowsy driving or employment that requires routine operation of transportation vehicles (e.g., truck/taxi driver, airline pilot) or hazardous equipment.
* Known allergy, hypersensitivity or contraindication to study medication
* Females: pregnant or nursing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2009-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Todd Arnedt, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Arnedt JT, Swanson LM, Dopp RR, Bertram HS, Mooney AJ, Huntley ED, Hoffmann RF, Armitage R. Effects of Restricted Time in Bed on Antidepressant Treatment Response: A Randomized Controlled Trial. J Clin Psychiatry. 2016 Oct;77(10):e1218-e1225. doi: 10.4088/JCP.15m09879. PMID 27529765

RESULTS

PARTICIPANT FLOW:
Groups:
- No Sleep Deprivation: 8 hours time in bed for two weeks plus fluoxetine for 8 weeks
- Late Bedtime Sleep Deprivation: 6 hours time in bed for two weeks plus fluoxetine for 8 weeks. Bedtime delayed by 2 hours.
- Early Risetime Sleep Deprivation: 6 hours time in bed for two weeks plus fluoxetine for 8 weeks. Rise time advanced by 2 hours.
Period: Overall Study
Arm/Group | No Sleep Deprivation | Late Bedtime Sleep Deprivation | Early Risetime Sleep Deprivation
Started | 19 | 24 | 25
Completed | 16 | 17 | 21
Not Completed | 3 | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- No Sleep Deprivation: 8 hours time in bed plus medication
  Sleep scheduling: 8 hours time in bed for two weeks
  Fluoxetine: 20-40 mg fluoxetine daily for 8 weeks
- Late Bedtime Sleep Deprivation: 6 hours time in bed plus medication
  Sleep scheduling:6 hours time in bed for two weeks; bedtime delayed by 2 hours
  Fluoxetine: 20-40 mg fluoxetine daily for 8 weeks
- Early Risetime Sleep Deprivation: 6 hours time in bed plus medication
  Sleep scheduling:6 hours time in bed for two weeks; risetime advanced by 2 hours
  Fluoxetine: 20-40 mg fluoxetine daily for 8 weeks
- Total: Total of all reporting groups
Arm/Group | No Sleep Deprivation | Late Bedtime Sleep Deprivation | Early Risetime Sleep Deprivation | Total
Number analyzed (Participants) | 19 | 24 | 25 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.4 (7.4) | 24.4 (5.6) | 25.7 (7.0) | 25.4 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 13 | 14 | 34
  Male | 12 | 11 | 11 | 34

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Rating Scale for Depression-17 Item Minus Sleep Items
Description: Total score on a clinician-rated measure of depressive symptoms, minus 3 sleep items Total score range: 0-46. Higher scores represent more severe depression.
Time Frame: Post-treatment (8 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- No Sleep Deprivation: 8 hours time in bed plus medication
  Sleep scheduling: 8 hours time in bed for 2 weeks
  Fluoxetine: 20-40 mg fluoxetine daily for 8 weeks
- Late Bedtime Sleep Deprivation: 6 hours time in bed plus medication
  Sleep scheduling: 6 hours time in bed for two weeks, with 2 hour delay in bedtime
  Fluoxetine: 20-40 mg fluoxetine daily for 8 weeks
- Early Risetime Sleep Deprivation: 6 hours time in bed plus medication
  Sleep scheduling: 6 hours time in bed for two weeks, with 2 hour advance in risetime
  Fluoxetine: 20-40 mg fluoxetine daily for 8 weeks
Arm/Group | No Sleep Deprivation | Late Bedtime Sleep Deprivation | Early Risetime Sleep Deprivation
Number analyzed (Participants) | 19 | 24 | 25
units on a scale | 6.1 (6.7) | 8.1 (4.4) | 6.3 (4.9)
Statistical Analysis 1: Comparison: No Sleep Deprivation vs Late Bedtime Sleep Deprivation vs Early Risetime Sleep Deprivation; Test type: Superiority or Other; p = .202, Mixed Models Analysis

2. Secondary Outcome: Quick Inventory of Depressive Symptoms (QIDS)
Description: Patient-reported depression symptom severity at post-treatment, total score. Total scores range from 0 to 27. Higher scores represent more severe depression.
Time Frame: Post-treatment (8 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- No Sleep Deprivation: 8 hours time in bed plus medication
  Sleep scheduling: 8 hours vs. 6 hours time in bed for two weeks
  Fluoxetine: 20-40 mg fluoxetine daily for 8 weeks
- Late Bedtime Sleep Deprivation: 6 hours time in bed plus medication
  Sleep scheduling: 6 hours time in bed for two weeks, with 2 hour delay of bedtime
  Fluoxetine: 20-40 mg fluoxetine daily for 8 weeks
- Early Risetime Sleep Deprivation: 6 hours time in bed plus medication
  Sleep scheduling: 6 hours time in bed for two weeks, with 2 hour advance of risetime
  Fluoxetine: 20-40 mg fluoxetine daily for 8 weeks
Arm/Group | No Sleep Deprivation | Late Bedtime Sleep Deprivation | Early Risetime Sleep Deprivation
Number analyzed (Participants) | 19 | 24 | 25
units on a scale | 5.3 (4.7) | 6.9 (3.3) | 6.7 (4.5)

3. Secondary Outcome: Pittsburgh Sleep Quality Index
Description: Self-report measure of sleep quality. The Pittsburgh Sleep Quality Index is a validated scale which measures self-reported sleep quality based on a wide variety of questions (duration, quality, disturbances, medication, etc.) and converts them to a scale which ranges from 0 to 21 where 6 or higher denotes poor sleep quality.
Time Frame: Baseline, 2 weeks and 8 weeks post-treatment
Population: At some time points, some participants did not show up to appointments or allow a particular test to be employed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | No Sleep Deprivation | Late Bedtime Sleep Deprivation | Early Risetime Sleep Deprivation
Number analyzed (Participants) | 14 | 14 | 15
units on a scale
  Baseline: number analyzed (Participants) | 10 | 12 | 13
  Baseline | 6.00 (2.828) | 8.67 (2.839) | 6.85 (3.236)
  Week 2: number analyzed (Participants) | 13 | 14 | 14
  Week 2 | 5.23 (2.204) | 6.07 (2.615) | 5.50 (2.312)
  Week 8: number analyzed (Participants) | 14 | 13 | 15
  Week 8 | 4.86 (2.248) | 6.23 (2.713) | 6.33 (2.944)

4. Secondary Outcome: Change in EEG Sleep Measures I: Total Sleep Time
Description: Measurement of EEG activity during sleep using polysomnography: Total Sleep Time is the length of time from sleep onset to final wake up minus any wakefulness during the night. It reflects the total amount of time asleep during the night.
Time Frame: Baseline, 2 weeks, 8 weeks
Population: Number of participants analyzed decreases in subsequent rows, as some participants dropped out or had unusable data.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | No Sleep Deprivation | Late Bedtime Sleep Deprivation | Early Risetime Sleep Deprivation
Number analyzed (Participants) | 19 | 24 | 25
minutes
  Baseline | 430.132 (60.9230) | 439.208 (36.3375) | 444.040 (19.7283)
  Week 2: number analyzed (Participants) | 17 | 18 | 22
  Week 2 | 435.382 (25.7206) | 337.75 (24.69) | 332.909 (17.0480)
  Week 8: number analyzed (Participants) | 15 | 17 | 21
  Week 8 | 439.6 (19.5231) | 428.264 (54.4570) | 433.333 (35.0347)

5. Secondary Outcome: Change in EEG Sleep Measures II (Sleep Efficiency)
Description: Measurement of EEG activity during sleep using polysomnography: Sleep efficiency [(total sleep time/time in bed)*100]
Time Frame: Baseline, 2 weeks, 8 weeks
Population: Subsequent rows have lower numbers of participants analyzed due to participant flow and/or unusable data.
Measure: Mean (Standard Deviation); unit: percent of sleep time
Arm/Group | No Sleep Deprivation | Late Bedtime Sleep Deprivation | Early Risetime Sleep Deprivation
Number analyzed (Participants) | 19 | 24 | 25
percent of sleep time
  Baseline | 89.7005 (12.62820) | 91.6829 (7.58117) | 92.8248 (4.01214)
  Week 2: number analyzed (Participants) | 17 | 18 | 22
  Week 2 | 90.7824 (5.29745) | 93.3322 (4.97614) | 92.9082 (4.01214)
  Week 8: number analyzed (Participants) | 15 | 17 | 21
  Week 8 | 91.6153 (4.03518) | 88.9224 (11.09279) | 90.3838 (7.17430)

6. Secondary Outcome: Change in Neuropsychological Functioning: Memory
Description: Change in different aspects of thinking (e.g., memory, attention, executive functioning)
Time Frame: Baseline, 2 weeks, 8 weeks
Population: At some time points, some participants did not show up to appointments or allow a particular test to be employed.
Measure: Mean (Standard Deviation); unit: words
Arm/Group | No Sleep Deprivation | Late Bedtime Sleep Deprivation | Early Risetime Sleep Deprivation
Number analyzed (Participants) | 17 | 17 | 21
words
  Baseline: number analyzed (Participants) | 17 | 16 | 21
  Baseline | 77.118 (17.1569) | 74.938 (10.2337) | 76.095 (13.4458)
  Week 2: number analyzed (Participants) | 17 | 17 | 20
  Week 2 | 76.647 (15.0829) | 81.529 (10.1311) | 77.400 (13.8579)
  Week 8: number analyzed (Participants) | 13 | 15 | 15
  Week 8 | 73.923 (12.1481) | 79.733 (7.4399) | 81.200 (14.1885)

7. Secondary Outcome: Change in Neurologic Functioning: Reaction Time
Description: Reaction Time is measured using a modified Go/No-go test of inhibitory control
Time Frame: 0, 2, 8 weeks
Population: At some time points, some participants did not show up to appointments or allow a particular test to be employed.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | No Sleep Deprivation | Late Bedtime Sleep Deprivation | Early Risetime Sleep Deprivation
Number analyzed (Participants) | 17 | 17 | 21
milliseconds
  Week 0 (Baseline): number analyzed (Participants) | 17 | 16 | 21
  Week 0 (Baseline) | 499.1545 (65.66508) | 528.3513 (135.86747) | 470.2942 (61.65017)
  Week 2: number analyzed (Participants) | 17 | 17 | 20
  Week 2 | 493.2579 (58.64806) | 519.8196 (60.68815) | 472.7244 (56.51599)
  Week 8: number analyzed (Participants) | 13 | 15 | 21
  Week 8 | 483.7349 (55.33537) | 557.1635 (188.22995) | 500.1197 (148.46524)

8. Secondary Outcome: Neurological Function (Emotional Perception)
Description: Emotional Perception is measured based on the percent of faces whose emotions are correctly identified using the Facial Emotion Perception Test (FEPT)
Time Frame: 0 weeks, 2 weeks, 8 weeks
Population: At some time points, some participants did not show up to appointments or allow a particular test to be employed.
Measure: Mean (Standard Deviation); unit: percentage of emotions accurately ID'ed
Arm/Group | No Sleep Deprivation | Late Bedtime Sleep Deprivation | Early Risetime Sleep Deprivation
Number analyzed (Participants) | 17 | 17 | 21
percentage of emotions accurately ID'ed
  0 weeks (Baseline): number analyzed (Participants) | 17 | 15 | 21
  0 weeks (Baseline) | 83.54 (10.549) | 86.24 (6.721) | 88.83 (7.321)
  Week 2 | 83.08 (6.938) | 88.15 (6.159) | 88.75 (7.099)
  Week 8: number analyzed (Participants) | 12 | 15 | 21
  Week 8 | 85.95 (8.585) | 89.15 (4.724) | 87.74 (4.708)

ADVERSE EVENTS:
Description: Adverse events judged to be related to the study and of moderate or greater severity
Groups:
- Late Bedtime Sleep Deprivation: 6 hours time in bed plus medication
  Sleep scheduling: 6 hours time in bed for two weeks, two hour delay of bedtime
  Fluoxetine: 20-40 mg fluoxetine daily for 8 weeks
- Early Risetime Sleep Deprivation: 6 hours time in bed plus medication
  Sleep scheduling: 6 hours time in bed for two weeks, two hour advance of risetime
  Fluoxetine: 20-40 mg fluoxetine daily for 8 weeks
Arm/Group | No Sleep Deprivation | Late Bedtime Sleep Deprivation | Early Risetime Sleep Deprivation
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 0/19 | 5/24 | 0/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Sleep Deprivation (N=19) | Late Bedtime Sleep Deprivation (N=24) | Early Risetime Sleep Deprivation (N=25)
Medication side effects (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) — Medication side effects judged to be moderately severe
Mood worsening (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Sample is largely young, healthy adults

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No